CLINICAL TRIAL: NCT05241886
Title: Evaluation Of Sarcopenia By Adding Anthropometric Measurements To The SARC-F Questionnaire
Brief Title: Evaluation of Sarcopenia With SARC-F and Anthropometric Measurement
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, Principal investigator, Ege University
Other Study IDs: Sarcopenia001
Record Dates: First submitted 2022-02-06; First posted 2022-02-16 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Sarcopenia; Older People
Keywords: Sarcopenia; SARC-F; Calf circumference; Mid upper arm circumference; EWGSOP; EWGSOP 2
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anthoropometric measurement, SARC- F questionnare — SARC-F, CC, MUAC

SUMMARY:
The aim of this study is to examine the performance of determining the sarcopenia by anthropometric measurements (mid-upper arm circumference and calf circumference) added to the SARC-F questionnaire developed as a screening tool for the risk of sarcopenia in the community-dwelling older adults. The risk of sarcopenia of the individuals over 65 years of age who applied to the Geriatrics Department of Ege University Medical Faculty Hospital Internal Diseases Department. was determined by the SARC-F questionnaire, muscle mass was established by bioelectrical impedance analysis, muscle strength was assessed by handgrip strength, physical performance was assessed by a 4-meter walking test and presence of malnutrition was assessed with an MNA-long form. For the diagnosis of sarcopenia; old (EWGSOP 1) and revised (EWGSOP 2) diagnostic criteria of Sarcopenia Study Group in Elderly Individuals of the European Union Geriatric Medicine Association were used. New parameters were obtained by adding calf circumference (SARC-CC) and mid-upper arm circumference (SARC-MUAC) measurements were added separately and together (SARC-CC-MUAC) to the SARC-F. For the calf circumference cut-off points of <31 cm and <33 cm and for the mid-upper arm circumference cut-off points of <25 cm and <31 cm were used for the sensitivity and specificity analyses.

DETAILED DESCRIPTION:
The population of the research is individuals aged 65 and over who applied to Ege University Medical Faculty Hospital Internal Diseases Department, Geriatrics BD Outpatient Clinic. For statistical power analysis; When α=0.05 and the power of the study are 0.80, the minimum number of samples required for the study was determined as 190. The relevant sample size was calculated with the G-Power 3.0.8 package program.

Data collection tools:

1. General information collection form: Investigator collect data about age, gender, chronic diseases, economic status, etc of participants
2. Measurement of Muscle Mass, Muscle Strength, and Gait Speed Body composition analysis was determined by electrical bioimpedance using the Tanita MC-780 multi-frequency segmental Body Composition Analyzer (Tanita Corporation, Tokyo). The appendicular skeletal muscle mass (ASM) was calculated with the Janssen equation for EWGSOP criteria and Sergi equation for EWGSOP 2 criteria. The appendicular muscle mass index (ASMI) was calculated based on the equation: ASM(kg) /height (m2).

   Muscle strength (kg) was assessed with the Takei Grip Strength Dynamometer®. Handgrip strength (HS) measurements were made with the subjects in a sitting position, with the elbow and wrist in full extension, three times with an interval of five seconds on both hands, and the highest value among the measurement results was used for analysis. Gender-specific cut-offs were used to define low muscle strength (30 and 20 kg in males and females) for EWGSOP criteria, and (27 and 16 kg in males and females) for EWGSOP 2 criteria. Usual gait speed (m/s) was performed by the subjects walking 4 m with usual speed and ≤0.8 m/s was defined as low walking speed.
3. Anthropometric measurement:

   In all participants, height was measured using a stadiometer to the nearest 0.1 cm, weight was measured unclothed to the nearest 0.1 kg using a calibrated balance scale. Body mass index (BMI) was calculated by the weight (kg)/height (m2) equation.

   The calf circumference (CC) of participants was measured with an inflexible tape measure, in the sitting position, with the knee flexed to 90º, and the circumference of the widest part of the calf. Both the standard CC cut-off (<31 cm) and population-specific cut-off (<33 cm) were used and compared in SARC-CalF analysis. Mid upper arm circumference (MUAC) was measured in a stand position, the mid-point of the participant's left upper arm- located between the acromion and olecranon- was marked when the elbow bent to a 90o angle and measured with the inflexible tape around the marked midpoint with the participant's arm hung down naturally.
4. Screening of sarcopenia risk and assessment of sarcopenia SARC-F, SARC-CalF, and SARC-MUAC were used for screening sarcopenia risk. For the SARC-F total score of ≥4, SARC-CalF ≥11, and SARC-MUAC≥11 were defined as positive sarcopenia risk. Investigator used EWGSOP and EWGSOP 2 criteria for sarcopenia diagnosis.
5. Statistic analysis: SPSS 25.0 (SPSS Statistics; IBM, Armonk, NY) and MedCalc Statistical Software 19.1.6-free trial (MedCalc Software, Ostend, Belgium) statistical package programs were used for statistical analysis. The level of significance was defined as p<0.05.

For categorical variables, the data were presented as numbers (percentage). Continuous variables with normal or skewed distribution were presented as mean (standard deviation) or median (interquartile range), respectively. Group differences were investigated using the t-test for normally distributed data and the Mann-Whitney test for skewed data and the X2 or Fisher's exact test for categorical data was used. Using EWGSOP and EWGSOP 2 criteria as the reference standard, the investigator calculated the diagnostic value of the SARC-F, SARC-CalF- 31, and SARC-CalF-33 [sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy] for identifying sarcopenia. A receiver operating characteristics (ROC) curve was used to compare the overall accuracy of SARC-F, SARC-CalF-31, and SARC-CalF-33. The area under the ROC curve (AUC) and 95% confidence interval (CI) were calculated.

The exclusion criteria are as follows: an implanted pacemaker, severe mental illness, unable to walk, severe heart failure, severe renal failure, clinically visible edema, and unable to communicate.

Participants in which all the evaluations in the research protocol were carried out and answered all the questions.

ELIGIBILITY:
Inclusion Criteria:

participants who applied to the geriatrics outpatient clinic for any reason

Exclusion Criteria:

Participants with an implanted pacemaker, severe mental illness, unable to walk, severe heart failure, severe renal failure, clinically visible edema, and unable to communicate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling participants aged 65 and over who applied to the geriatrics outpatient clinic for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
sarcopenia prevalance | Day 1
  number
SARC-F score | Day 1
  number
mid-upper arm circumference | Day 1
  cm
calf circumference | Day 1
  cm
Appendicular skeletal muscle mass index | Day 1
  kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: yasemin A Atik-Altinok, PhD, Principal Investigator — Ege University; Devrim Bozkurt, Assoc Prof, Study Director — Ege University; Sumru Savaş, Assoc Prof, Principal Investigator — Ege University; Reci Meseri, Assoc Prof, Principal Investigator — Ege University; Fulden Saraç, Prof Dr, Principal Investigator — Ege University; Fehmi Akçiçek, Prof Dr, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd-El-Gawad WM, Abou-Hashem RM, El Maraghy MO, Amin GE. The validity of Geriatric Nutrition Risk Index: simple tool for prediction of nutritional-related complication of hospitalized elderly patients. Comparison with Mini Nutritional Assessment. Clin Nutr. 2014 Dec;33(6):1108-16. doi: 10.1016/j.clnu.2013.12.005. Epub 2013 Dec 28. PMID 24418116
- [Background] Ates Bulut E, Soysal P, Dokuzlar O, Kocyigit SE, Aydin AE, Yavuz I, Isik AT. Validation of population-based cutoffs for low muscle mass and strength in a population of Turkish elderly adults. Aging Clin Exp Res. 2020 Sep;32(9):1749-1755. doi: 10.1007/s40520-019-01448-4. Epub 2020 Jan 2. PMID 31898170
- [Background] Bahat G, Yilmaz O, Kilic C, Oren MM, Karan MA. Performance of SARC-F in Regard to Sarcopenia Definitions, Muscle Mass and Functional Measures. J Nutr Health Aging. 2018;22(8):898-903. doi: 10.1007/s12603-018-1067-8. PMID 30272090
- [Background] Fu X, Tian Z, Thapa S, Sun H, Wen S, Xiong H, Yu S. Comparing SARC-F with SARC-CalF for screening sarcopenia in advanced cancer patients. Clin Nutr. 2020 Nov;39(11):3337-3345. doi: 10.1016/j.clnu.2020.02.020. Epub 2020 Feb 22. PMID 32143888
- [Background] Sergi G, De Rui M, Veronese N, Bolzetta F, Berton L, Carraro S, Bano G, Coin A, Manzato E, Perissinotto E. Assessing appendicular skeletal muscle mass with bioelectrical impedance analysis in free-living Caucasian older adults. Clin Nutr. 2015 Aug;34(4):667-73. doi: 10.1016/j.clnu.2014.07.010. Epub 2014 Jul 24. PMID 25103151
- [Background] da Luz MCL, Pinho CPS, Bezerra GKA, da Conceicao Chaves de Lemos M, da Silva Diniz A, Cabral PC. SARC-F and SARC-CalF in screening for sarcopenia in older adults with Parkinson's disease. Exp Gerontol. 2021 Feb;144:111183. doi: 10.1016/j.exger.2020.111183. Epub 2020 Dec 3. PMID 33279661
- [Background] Hajaoui M, Locquet M, Beaudart C, Reginster JY, Petermans J, Bruyere O. Sarcopenia: Performance of the SARC-F Questionnaire According to the European Consensus Criteria, EWGSOP1 and EWGSOP2. J Am Med Dir Assoc. 2019 Sep;20(9):1182-1183. doi: 10.1016/j.jamda.2019.05.021. No abstract available. PMID 31455509
- [Background] Drey M, Ferrari U, Schraml M, Kemmler W, Schoene D, Franke A, Freiberger E, Kob R, Sieber C. German Version of SARC-F: Translation, Adaption, and Validation. J Am Med Dir Assoc. 2020 Jun;21(6):747-751.e1. doi: 10.1016/j.jamda.2019.12.011. Epub 2020 Jan 21. PMID 31980396